CLINICAL TRIAL: NCT02851719
Title: Outpatient Biofeedback in Addition to Home Pelvic Floor Muscle Training for Stress Urinary Incontinence: a Randomized Controlled Trial
Brief Title: Outpatient Biofeedback in Addition to Home Pelvic Floor Muscle Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fatima Fitz, Physical Therapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Pelvic Floor; Exercise; Patient Compliance
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity; Patient Compliance | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF group (Experimental): 24 outpatient sessions of the PFMT (twice a week) using manometric-based BF equipment and daily home PFMT exercises.
  Interventions: Other: PFMT with biofeedback + Home PFMT
- PFMT group (Active Comparator): 24 outpatient sessions (twice a week) of PFMT without BF and daily home PFMT exercises.
  Interventions: Other: PFMT without biofeedback + Home PFMT

INTERVENTIONS:
Other: PFMT with biofeedback + Home PFMT — 24 outpatient sessions PFMT with biofeedback (twice a week). Simultaneously, it was prescribed a home exercise daily program during three months (supervised treatment).
  Other Names: Biofeedback
  Arms: BF group
Other: PFMT without biofeedback + Home PFMT — 24 outpatient sessions PFMT without biofeedback (twice a week). Simultaneously, it was prescribed a home exercise daily program during three months (supervised treatment).
  Other Names: PFMT alone
  Arms: PFMT group

SUMMARY:
To test whether biofeedback (BF) added to pelvic floor muscle training (PFMT) promotes additional benefits over PFMT alone in the stress urinary incontinence (SUI) treatment.

DETAILED DESCRIPTION:
Introduction: The aim of this study was to test the hypothesis that outpatient BF added to home PFMT results in increased frequency of home exercises sets per month performed by the patients and objective cure rate after 3 months of supervised training. Secondarily, to investigate other subjective and objective clinical parameters in the groups that received or not BF together with PFMT after 3 months of supervised training, and in a longer term of 9-month follow-up.

Method: 72 incontinent women were randomized to the: BF Group (outpatient BF + home PFMT) or PFMT Group (outpatient PFMT + home PFMT).

Assessments: baseline after 3 months of supervised treatment and at 9-month follow-up (after 6 additional months of home PFMT without supervision).

Primary outcomes: adherence - monthly exercises sets performed (exercise diary) and objective cure of SUI (pad test) after 3 months.

Secondary outcomes: urinary symptoms, muscle function, quality of life, adhesion and subject cure at the two time-points.

ELIGIBILITY:
Inclusion Criteria:

* SUI and mixed urinary incontinence with predominant symptoms of SUI with ≥ 2 g of leakage measured by pad test

Exclusion Criteria:

* younger than 18 years old
* chronic degenerative diseases
* pelvic organ prolapse greater than stage I by POP-Q
* neurologic or psychiatric diseases
* previously undergone pelvic floor re-education programs and/or previous pelvic floor surgeries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in pad test | Baseline, after 3 months of supervised treatment and at 9-month follow-up
  To quantify the severity of SUI and as the tool to estimate objective cure rate

SECONDARY OUTCOMES:
Change in 7-Day Voiding Diary | Baseline, after 3 months of supervised treatment and at 9-month follow-up
  To assess the loss efforts
Change in pelvic floor muscle function (Oxford Grading Scale) | Baseline, after 3 months of supervised treatment and at 9-month follow-up
  To assess the function of the pelvic floor muscle
Change in pelvic floor muscle function (Peritron manometer) | Baseline, after 3 months of supervised treatment and at 9-month follow-up
  To assess the function of the pelvic floor muscle
Change in Incontinence Quality-of-Life Questionnaire (I-QoL) | Baseline, after 3 months of supervised treatment and at 9-month follow-up
  To quantify the impact of SUI on quality of life
Subjective cure of SUI ("satisfied" or "dissatisfied") | After 3 months of supervised treatment and at 9-month follow-up
  To evaluate the patient satisfaction with treatment
Frequency and adhesion to the home exercises | After 3 months of supervised treatment and at 9-month follow-up
  The weekly frequency (days/week that patients performed at least 1 set of exercises) and the number of sets per day
Frequency of the outpatient sessions | After 3 months of supervised treatment
  The frequency of the outpatient sessions was monitored

CONTACTS AND LOCATIONS:
Overall Officials: Fatima F Fitz, M.Sc, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) collected in this study are being analyzed by the researchers to be available.